CLINICAL TRIAL: NCT04427098
Title: Intermediate Dose Enoxaparin in Hospitalized Patients With Moderate-severe COVID19: A Pilot Phase II Single-arm Study, INHIXACOVID19
Brief Title: Enoxaparin in COVID-19 Moderate to Severe Hospitalized Patients
Acronym: INHIXACOV19
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Pierluigi Viale, Professor of Infectious Diseases, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-001308-40
Record Dates: First submitted 2020-05-29; First posted 2020-06-11 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-08

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Enoxaparin

STUDY DESIGN:
Intervention Model Description: The study consists of two parts:
  * a phase II single-arm interventional prospective study including all patients treated with the study drug;
  * an observational prospective cohort study including all patients screened for receiving the study drug but not included in the phase II study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- a phase II single-arm interventional prospective study (Active Comparator): Patients included in the interventional study will receive subcutaneous enoxaparin in a single daily dose of:
  * 60 mg once daily in case of body weight of 45 to 60 kg
  * 80 mg per day in case of weight from 61 to 100 kg or
  * 100 mg once daily in case of bodyweight >100 kg
  Enoxaparin will be started on the first day of COVID19 diagnosis and continued for 14 days.
  Interventions: Drug: Enoxaparin 40 Mg/0.4 mL Injectable Solution
- observational cohort study (Experimental): Patients included in the observational cohort will will receive standard thrombo-prophylaxis with subcutaneous enoxaparin 40 mg/die
  Interventions: Drug: Enoxaparin

INTERVENTIONS:
Drug: Enoxaparin 40 Mg/0.4 mL Injectable Solution — Subcutaneous enoxaparin 40 mg once daily for 14 days.
  Other Names: INHIXA 4,000 UI (40 mg) / 0.4 ml
  Arms: a phase II single-arm interventional prospective study
Drug: Enoxaparin — Subcutaneous enoxaparin for 14 days: 60 mg once daily in case of body weight of 45 to 60 kg; 80 mg once daily in case of weight from 61 to 100 kg; 100 mg once daily in case of bodyweight >100 kg
  Other Names: INHIXA 6,000 UI (60 mg) / 0.6 ml; INHIXA 8,000 UI (80 mg) / 0.8 ml; INHIXA 10,000 UI (100 mg)/ 1 ml
  Arms: observational cohort study

SUMMARY:
General objective of the study To assess the efficacy and safety of enoxaparin in hospitalized patients with moderate to severe COVID-19 (Coronavirus Disease 2019) infection.

Study Design

The study consists of two parts:

* a phase II single-arm interventional prospective study including all patients treated with the study drug;
* an observational prospective cohort study including all patients screened for receiving the study drug but not included in the phase II study.

Patients will be enrolled from "date of study approval" for 1 month. Each patient will be followed-up for a minimum of 90 days after COVID19 diagnosis.

DETAILED DESCRIPTION:
General objective of the study To assess the efficacy and safety of enoxaparin in hospitalized patients with moderate to severe COVID-19 infection.

Specific objectives Primary Endpoints To investigate the efficacy of enoxaparin in improving the clinical outcome of hospitalized patients with moderate to severe COVID-19.

* All-cause in-hospital, 30-day and 90-day mortality rates.
* Evolution of the clinical severity during treatment.
* ICU admission and length of ICU stay.
* Length of hospital stay.

Secondary Endpoints To analyse the safety of enoxaparin in hospitalized patients with with moderate to severe COVID-19.

* Rate of adverse events (AEs) during treatment, at the end of treatment (EOT) and at 30 days after EOT.
* Severity of AEs classified according to common terminology criteria for adverse events (CTCAE). The worst degree ever suffered will be considered.

To describe the rates and the types of thromboembolic events among hospitalized patients with confirmed diagnosis of COVID-19.

* Occurrence of thromboembolic event at 90 days after COVID-19 diagnosis.
* Description of the type, distribution and severity of thromboembolic events.

Study Design Overall Design

The study consists of two parts:

* a phase II single-arm interventional prospective study including all patients treated with the study drug;
* an observational prospective cohort study including all patients screened for receiving the study drug but not included in the phase II study.

Patients will be enrolled from "date of study approval" for 1 month. Each patient will be followed-up for a minimum of 90 days after COVID19 diagnosis.

End of Study Definition A participant is considered to have completed the study if he/she has completed the last scheduled procedure shown in the Schedule of assessments. The end of the study is defined as the date of the last scheduled procedure shown in the Schedule of assessments for the last participant in the trial.

Study Population

Definitions

Clinical severity of COVID-19 will be assessed at the diagnosis of COVID19, during the treatment with the study drug, and at the end of treatment according to the following criteria (1):

* Mild patients: only show mild symptoms without radiographic features
* Moderate patients: have fever, respiratory symptoms, and radiographic signs of pneumonia
* Severe patients: have fever, respiratory symptoms, and radiographic signs of pneumonia plus at least one of three criteria: (1) RR (respiratory rate) >30 times/min, (2) oxygen saturation <93% on ambient air, (3) PaO2/FiO2 (Oxygen partial pressure/inspired oxygen fraction ) <300 mmHg.
* Critical patients: meet one of three criteria: (1) respiratory failure needing invasive ventilation, (2) septic shock, (3) multiple organ failure.

Major bleeding will be defined according to the ISTH (International Society of Thrombosis and Haemostasis) criteria as one of the following:

* Fatal bleeding
* Symptomatic bleeding in a critical area or organ, such as intracranial, intraspinal, intraocular, retroperitoneal, intra-articular or pericardial, or intramuscular with compartment syndrome
* Bleeding causing a fall in haemoglobin level of 2 g/dL or more, or leading to transfusion of two or more units of whole blood or red cells (11).

Treatments Administration and monitoring of study drug

All patients screened for being included in the study will receive standard thrombo-prophylaxis with LMWH (low molecular weight heparin) (e.g. enoxaparin 40 mg/die). Patients included in the observational cohort will continue on standard thrombo-prophylaxis, while patients included in the interventional study will receive subcutaneous enoxaparin in a single daily dose of:

* 60 mg once daily in case of body weight of 45 to 60 kg
* 80 mg per day in case of weight from 61 to 100 kg or
* 100 mg once daily in case of bodyweight >100 kg Enoxaparin will be started on the first day of COVID19 diagnosis and continued for 14 days, after determination of baseline PT (prothrombin time), aPTT (activated partial thromboplastin time), complete blood cell count and creatinine levels.

After reaching the steady state (usually after the third dose), heparin levels will be measured with the determination of anti-Xa activity on a blood sample obtained at 4 hours after the morning injection. LMWH dose may be then increased or reduced on the basis of target anti-Xa activity (0.4-0.6 antiFXa (Anti Factor X activated) UI/ml (International Unit/ml) for intermediate doses). The determination of anti-Xa activity will be repeated on the fifth or sixth day to monitor any drug accumulation.

Complete blood cell count will be obtained every second day to monitor for heparin induced thrombocytopenia.

Single low dose antiplatelet agents will be allowed. In all patients, RT-PCR (reverse transcription-polymerase chain reaction) nasopharyngeal swabs will be performed every 7 days to assess virus clearance and blood samples will be collected at baseline and on day 7 and will be retrospectively analysed to measure viral load.

Follow up procedures Patients will be followed-up to 90 days after study drug initiation. Follow-up information will be collected via telephone calls, patient medical records and/or clinical visits according to clinical evolution.

This is a pilot study and an initial sample of 100 patients for the phase II single-arm interventional trial is established. Even if currently precise data are not available, it can be assumed that the composite endpoint is around 30% in patient treated with the standard thromboprophylaxis dose of enoxaparin. To verify the hypothesis that the experimental treatment may produce a halving of this endpoint (from 30% to 15%), 300 patients (200 for the observational cohort and 100 for the phase II cohort; ratio 2:1) are needed with a 80% power and a 0,05 bilateral alpha error. As stated above a first safety analysis after enrolling the first 50 patients in the interventional study arm is planned and it will be done by an independent committee. According to safety and efficacy data obtained, using as control the observational cohort, a large study with a more robust design is planned.

ELIGIBILITY:
Inclusion Criteria:

* For both interventional study and observational cohort, hospitalized patients are eligible to be included if the following criteria apply:

Inclusion criteria:

* Age >=18 y
* Microbiologically confirmed COVID-19 infection
* Patients with moderate to severe disease according to study definitions (see below)
* Informed consent to participate and to use data for interventional study, only to use data for observational cohort

Exclusion Criteria:

* Participants are excluded from the interventional study if any of the following criteria apply:

  * Thrombocytopenia (platelet count < 50.000 mm3)
  * Coagulopathy: INR (International normalized ratio) >1.5, aPTT ratio >1.4
  * Impaired renal function (clearance to creatinine less than 15 ml/min)
  * Known hypersensitivity to heparin
  * History of heparin induced thrombocytopenia
  * Presence of an active bleeding or a pathology susceptible of bleeding in presence of anticoagulation (e.g. recent haemorrhagic stroke, peptic ulcer, malignant tumors at hig risk of haemorrhages, recent neurosurgery or ophthalmic surgery, vascular aneurysms, arteriovenous malformations)
  * Body weight <45 or > 150 kg
  * Concomitant anticoagulant treatment for other indications ( eg atrial fibrillation, venous thromboembolism , prosthetic heart valves).
  * Dual antiplatelet therapy
  * Pregnant or breast-feeding women

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 301 (Actual)
Dates: Start 2020-05-22 (Actual); Primary Completion 2021-09-29 (Actual); Study Completion 2021-09-29 (Actual)

PRIMARY OUTCOMES:
Mortality | 30 days and 90 days from the first LMWH subcutaneous injection
  Rates of hospitalized patients dead for all-cause within 30 days and 90 days from the first LMWH subcutaneous injection
Effectivness of enoxaparin on the outcome of COVID 19. | This evaluation will be performed at 30 days and 90 days from the first LMWH subcutaneous injection
  Based on the four levels scale of severity of symptoms. Any change from one level to another will be detected for all the enrolled patients.
ICU admission and length of ICU stay | This evaluation will be performed at 14 days (the last day of treatment adminstration), at 30 days and 90 days from the first LMWH subcutaneous injection
  Evolution of the clinical severity during treatment, based on the number and rate of patients admitted to ICU and the length of their ICU stay
Lenght of hospital stay | This evaluation will be performed at 90 days from admission
  Difference between groups in number of days of hospitalization from admission to discharge

SECONDARY OUTCOMES:
To describe the rates and the types of thromboembolic events among hospitalized patients with confirmed diagnosis of COVID-19. | 90 days
  Occurrence of thromboembolic event at 90 days after COVID-19 diagnosis. Description of the type, distribution and severity of thromboembolic events.
Advers Events | 45 days
  Rate of adverse events (AEs) during treatment, at the end of treatment (EOT) and at 30 days after EOT.
  • Severity of AEs classified according to common terminology criteria for adverse events (CTCAE). The worst degree ever suffered will be considered.

CONTACTS AND LOCATIONS:
Overall Officials: Pierluigi Viale, MD, Principal Investigator — Infectious Diseases Unit, Dep. Med. and Surg. Science University of Bologna
Locations (13):
- Italy (13):
  - Policlinico S. Orsola Malpighi Dipartimento Malattie Infettive, Bologna, Emilia-Romagna
  - Azienda Ospedaliero-Universitaria di Parma Anestesia e Rianimazione Dipartimento di Medicina e Chirurgia, Parma, Emilia-Romagna
  - I.R.C.C.S. "Casa Sollievo della Sofferenza", San Giovanni Rotondo (FG) UOVD Emostasi e trombosi- Poliambulatorio Giovanni Paolo II Viale Padre Pio n.7 San Giovanni Rotondo (FG), San Giovanni Rotondo, Foggia
  - Fondazione Poliambulanza Chirurgia Vascolare, Brescia
  - Piazzale Spedali Civili, 1, 25123 Brescia BS Medicina Interna UniBS 2° Medicina ASST Spedali Civili, Brescia
  - Azienda Ospedaliero-Universitaria "Policlinico - V. Emanuele", Catania Anestesia e Rianimazione UO Malattie Infettive, Catania
  - ASST Cremona Unità Operativa di Chirurgia Vascolare Dipartimento di Medicina di Laboratorio e di Radiologia- Centro Emostasi e Trombosi, Cremona
  - Ospedale Morgagni Pierantoni U.O.C. Malattie Infettive, Forlì
  - Ospedale Carlo Poma di Mantova MALATTIE INFETTIVE Padiglione 37 Str. Lago Paiolo, 10, 46100 Mantova, Mantova
  - AZIENDA OSPEDALIERA Regionale S CARLO POTENZA Struttura Complessa Interaziendale "Malattie Infettive", Matera
  - Ospedale San Raffaele Unità Funzionale dell'Unità Operativa di Malattie Infettive Osp. San Raffaele, Milan
  - Ospedale Amedeo di Savoia Torino Università di Torino Malattie Infettive, Torino
  - Azienda Ospedaliera Universitaria Integrata Verona UOC Malattie Infettive e Tropicali, Verona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cosmi B, Giannella M, Fornaro G, Cristini F, Patacca A, Castagna A, Mazzaferri F, Testa S, Pan A, Lupi M, Brambilla P, Montineri A, Frattima S, Bignami EG, Salvetti M, De Stefano G, Grandone E, Di Perri G, Rozzini R, Stella A, Romagnoli A, Drago F, Viale P. Intermediate dose enoxaparin in hospitalized patients with moderate-severe COVID-19: a pilot phase II single-arm study, INHIXACOVID19. BMC Infect Dis. 2023 Oct 24;23(1):718. doi: 10.1186/s12879-023-08297-7. PMID 37875792